CLINICAL TRIAL: NCT02504320
Title: A Phase 1, Randomized, Open-Label, Single-Dose, 4-Way Crossover Study to Assess the Relative Bioavailability of Four 80 mg Febuxostat XR Formulations
Brief Title: Phase 1, Febuxostat XR Relative Bioavailability Study
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Takeda (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Basic Science
Other Study IDs: Febuxostat XR-1011; U1111-1168-1117 (Other: WHO)
Record Dates: First submitted 2015-07-20; First posted 2015-07-21 (Estimated); Results first posted 2017-01-19 (Estimated); Last update posted 2017-01-19 (Estimated); Status verified 2016-11

CONDITIONS: Healthy Volunteers
Keywords: Drug therapy
MeSH Terms: interventions — F 4

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (4):
- Treatment Sequence ABDC (Experimental): Febuxostat XR 80 mg capsule Formulation 1 (F1), orally, once on Day 1 of Period 1 (A), followed by at least a 7-day washout period, followed by Febuxostat XR 80 mg capsule Formulation 2 (F2), orally, once on Day 1 of Period 2 (B), followed by at least a 7-day washout period, followed by Febuxostat XR 80 mg capsule Formulation 4 (F4), orally, once on Day 1 of Period 3 (D), followed by at least a 7-day washout period, followed by Febuxostat XR 80 mg capsule Formulation 3 (F3), orally, once on Day 1 of Period 4 (C).
  Interventions: Drug: Febuxostat XR 80 mg Capsule F1; Drug: Febuxostat XR 80 mg Capsule F2; Drug: Febuxostat XR 80 mg Capsule F3; Drug: Febuxostat XR 80 mg Capsule F4
- Treatment Sequence DACB (Experimental): Febuxostat XR 80 mg capsule F4, orally, once on Day 1 of Period 1 (D), followed by at least a 7-day washout period, followed by Febuxostat XR 80 mg capsule F1 orally, once on Day 1 of Period 2 (A), followed by at least a 7-day washout period, followed by Febuxostat XR 80 mg capsule F3, orally, once on Day 1 of Period 3 (C), followed by at least a 7-day washout period, followed by Febuxostat XR 80 mg capsule F2, orally, once on Day 1 of Period 4 (B).
  Interventions: Drug: Febuxostat XR 80 mg Capsule F1; Drug: Febuxostat XR 80 mg Capsule F2; Drug: Febuxostat XR 80 mg Capsule F3; Drug: Febuxostat XR 80 mg Capsule F4
- Treatment Sequence CDBA (Experimental): Febuxostat XR 80 mg capsule F3, orally, once on Day 1 of Period 1 (C), followed by at least a 7-day washout period, followed by Febuxostat XR 80 mg capsule F4 orally, once on Day 1 of Period 2 (D), followed by at least a 7-day washout period, followed by Febuxostat XR 80 mg capsule F2, orally, once on Day 1 of Period 3 (B), followed by at least a 7-day washout period, followed by Febuxostat XR 80 mg capsule F1, orally, once on Day 1 of Period 4 (A).
  Interventions: Drug: Febuxostat XR 80 mg Capsule F1; Drug: Febuxostat XR 80 mg Capsule F2; Drug: Febuxostat XR 80 mg Capsule F3; Drug: Febuxostat XR 80 mg Capsule F4
- Treatment Sequence BCAD (Experimental): Febuxostat XR 80 mg capsule F2, orally, once on Day 1 of Period 1 (B), followed by at least a 7-day washout period, followed by Febuxostat XR 80 mg capsule F3 orally, once on Day 1 of Period 2 (C), followed by at least a 7-day washout period, followed by Febuxostat XR 80 mg capsule F1, orally, once on Day 1 of Period 3 (A), followed by at least a 7-day washout period, followed by Febuxostat XR 80 mg capsule F4, orally, once on Day 1 of Period 4 (D).
  Interventions: Drug: Febuxostat XR 80 mg Capsule F1; Drug: Febuxostat XR 80 mg Capsule F2; Drug: Febuxostat XR 80 mg Capsule F3; Drug: Febuxostat XR 80 mg Capsule F4

INTERVENTIONS:
Drug: Febuxostat XR 80 mg Capsule F1 — Febuxostat extended-release (XR) capsules formulation 1
Drug: Febuxostat XR 80 mg Capsule F2 — Febuxostat XR capsules formulation 2
Drug: Febuxostat XR 80 mg Capsule F3 — Febuxostat XR capsules formulation 3
Drug: Febuxostat XR 80 mg Capsule F4 — Febuxostat XR capsules formulation 4

SUMMARY:
This study will assess the relative bioavailability, safety and tolerability following administration of 80 mg single oral doses of 4 febuxostat extended release (XR) formulations.

DETAILED DESCRIPTION:
The drug being tested is this study is febuxostat XR. Four different formulations of febuxostat XR are being tested to see how the drug moves through the body. This study will look at safety and side effects in people who take febuxostat XR.

This cross-over study will enroll approximately 78 patients. Participants will be randomly assigned to 1of 4 sequences which will determine the order of the 4 treatments received:

* Febuxostat XR 80 mg capsule Formulation 1
* Febuxostat XR 80 mg capsule Formulation 2
* Febuxostat XR 80 mg capsule Formulation 3
* Febuxostat XR 80 mg capsule Formulation 4

Participants will take 1 dose on Day 1 with a washout period between each period.

This single-center trial will be conducted in the United States. The overall time to participate in this study is up to 80 days. Participants will make multiple visits to the clinic including a period of confinement, and will be contacted by telephone 30 days after last dose of study drug for a follow-up assessment.

ELIGIBILITY:
Inclusion Criteria:

1. In the opinion of the investigator, the participant is capable of understanding and complying with protocol requirements.
2. The participant or, when applicable, the participant's legally acceptable representative signs and dates a written, informed consent form and any required privacy authorization prior to the initiation of any study procedures including requesting that a participant fast for any laboratory evaluations.
3. Is a healthy male or female and aged 18 to 55 years, inclusive, at the time of informed consent and first study medication dose.
4. Weighs at least 50.0 kg and has a body mass index (BMI) from 18.0 to 30.0 kg/m2, inclusive at Screening.
5. A male participant who is nonsterilized and sexually active with a female partner of childbearing potential agrees to use adequate contraception from signing of informed consent throughout the duration of the study and for 30 days after the last dose.
6. A female participant of childbearing potential who is sexually active with a nonsterilized male partner agrees to use routinely adequate contraception from signing of informed consent,
7. Is willing to refrain from strenuous exercise from Day -1 of Period 1 until Study Exit (Day 3 of Period 4).
8. Has estimated glomerular filtration rate (eGFR) ≥90 mL/min at Screening and Check-in (Day -1 of Period 1).

Exclusion Criteria:

1. Has received any investigational compound within 30 days prior to the first dose of study medication.
2. Has received febuxostat in a previous clinical study or as a therapeutic agent.
3. Is an immediate family member, study site employee, or is in a dependant relationship with a study site employee who is involved in the conduct of this study.
4. Has uncontrolled, clinically significant (CS) disease or other abnormality, which may impact the ability of the participant to participate or potentially confound the study results.
5. Has a known hypersensitivity to any component of the formulation of XO inhibitors, xanthine compounds, caffeine, or any component of the formulation of febuxostat capsules.

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 78 (Actual)
Dates: Start 2015-08; Primary Completion 2015-09 (Actual); Study Completion 2015-10 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Medical Director Clinical Science, Study Director — Takeda
Locations (1):
- Austin, Texas, United States

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants took part in the study at 1 investigative site in the United States from 29 June 2015 to 01 October 2015.
Pre-assignment Details: Healthy participants were enrolled equally in 1 of 4 sequences which determined order of treatment: Regimen A (Febuxostat extended release [XR] 80 mg capsule [cap] Formulation [F] 1), B (Febuxostat XR 80 mg cap F2), C (Febuxostat XR 80 mg cap F3) and D (Febuxostat XR 80 mg cap F4). Each regimen is separated by a 7-day washout period.
Period: Treatment Period 1
Arm/Group | Treatment Sequence ABDC | Treatment Sequence DACB | Treatment Sequence CDBA | Treatment Sequence BCAD
Started | 19 | 19 | 20 | 20
Completed | 19 | 19 | 19 | 20
Not Completed | 0 | 0 | 1 | 0
Not completed — Positive Drug Screen | 0 | 0 | 1 | 0
Period: Treatment Period 2
Arm/Group | Treatment Sequence ABDC | Treatment Sequence DACB | Treatment Sequence CDBA | Treatment Sequence BCAD
Started | 19 | 19 | 19 | 20
Completed | 19 | 18 | 19 | 20
Not Completed | 0 | 1 | 0 | 0
Not completed — Positive Drug Screen | 0 | 1 | 0 | 0
Period: Treatment Period 3
Arm/Group | Treatment Sequence ABDC | Treatment Sequence DACB | Treatment Sequence CDBA | Treatment Sequence BCAD
Started | 19 | 18 | 19 | 20
Completed | 19 | 18 | 18 | 19
Not Completed | 0 | 0 | 1 | 1
Not completed — Positive Drug Screen | 0 | 0 | 0 | 1
Not completed — Adverse Event | 0 | 0 | 1 | 0
Period: Treatment Period 4
Arm/Group | Treatment Sequence ABDC | Treatment Sequence DACB | Treatment Sequence CDBA | Treatment Sequence BCAD
Started | 19 | 18 | 18 | 19
Completed | 19 | 18 | 18 | 19
Not Completed | 0 | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Population: Safety Set included all participants who were enrolled and received at least 1 dose of study drug.
Groups:
- Total: Total of all reporting groups
Arm/Group | Treatment Sequence ABDC | Treatment Sequence DACB | Treatment Sequence CDBA | Treatment Sequence BCAD | Total
Number analyzed (Participants) | 19 | 19 | 20 | 20 | 78
Age, Continuous [Mean (Standard Deviation); unit: years] | 31.7 (7.56) | 30.7 (6.51) | 34.0 (8.87) | 31.2 (7.78) | 31.9 (7.70)
Gender [Count of Participants; unit: Participants]
  Female | 10 | 10 | 9 | 14 | 43
  Male | 9 | 9 | 11 | 6 | 35
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Hispanic or Latino | 11 | 7 | 9 | 10 | 37
  Not Hispanic or Latino | 8 | 12 | 11 | 10 | 41
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Asian | 0 | 0 | 0 | 1 | 1
  Black or African American | 4 | 7 | 6 | 6 | 23
  White | 15 | 11 | 14 | 13 | 53
  Multiracial | 0 | 1 | 0 | 0 | 1
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 19 | 19 | 20 | 20 | 78
Height [Mean (Standard Deviation); unit: cm] | 167.6 (10.13) | 171.1 (11.75) | 167.5 (9.70) | 165.7 (6.67) | 167.9 (9.71)
Weight [Mean (Standard Deviation); unit: kg] | 72.98 (12.685) | 79.05 (11.846) | 71.22 (12.350) | 69.72 (11.015) | 73.17 (12.273)
Body Mass Index (BMI) [Mean (Standard Deviation); unit: kg/m^2] | 25.84 (2.663) | 26.98 (2.722) | 25.29 (3.168) | 25.28 (2.802) | 25.83 (2.878)
Smoking Classification [Count of Participants; unit: Participants]
  Has Never Smoked | 13 | 14 | 13 | 18 | 58
  Is a Current Smoker | 0 | 0 | 0 | 0 | 0
  Is an Ex-smoker | 6 | 5 | 7 | 2 | 20
Alcohol Classification [Count of Participants; unit: Participants]
  Has Never Drunk | 4 | 6 | 6 | 7 | 23
  Is a Current Drinker | 8 | 9 | 6 | 4 | 27
  Is an Ex-drinker | 7 | 4 | 8 | 9 | 28
Xanthine/Caffeine Consumption [Count of Participants; unit: Participants]
  Yes | 12 | 13 | 12 | 14 | 51
  No | 7 | 6 | 8 | 6 | 27
Female Reproductive Status [Count of Participants; unit: Participants]
  Not Applicable (Participant is Male) | 9 | 9 | 11 | 6 | 35
  Female of Childbearing Potential | 7 | 9 | 8 | 12 | 36
  Surgically Sterile | 2 | 1 | 0 | 2 | 5
  Postmenopausal | 1 | 0 | 1 | 0 | 2
Estimated Glomerular Filtration Rate (eGFR) [Mean (Standard Deviation); unit: mL/min] — eGFR is calculated using the Cockcroft-Gault formula.
  mL/min
    Screening (n=19, 19, 19, 20) | 111.42 (11.815) | 112.84 (11.987) | 108.05 (11.664) | 114.00 (13.377) | 111.61 (12.211)
    Check-in (n=19, 19, 20, 20) | 115.53 (12.294) | 115.26 (12.229) | 112.00 (10.964) | 116.55 (12.845) | 114.82 (11.987)

OUTCOME MEASURES:

1. Primary Outcome: Mean Cmax: Maximum Observed Plasma Concentration for Febuxostat
Description: Maximum observed plasma concentration (Cmax) is the peak plasma concentration of a drug after administration, obtained directly from the plasma concentration-time curve.
Time Frame: Day 1 pre-dose and at multiple time points (up to 48 hours) post-dose
Population: Participants with valid parameters for Regimen D and at least one of the test regimen were included in the analyses for this outcome measure. Here, number of participants analyzed is the participants who were evaluable for this outcome measure.
Measure: Mean (Standard Deviation); unit: ng/mL
Groups:
- Regimen A: Febuxostat XR 80 mg Formulation 1: Febuxostat XR 80 mg capsule formulation 1 (F1), orally, once on Day 1 of periods 1, 2, 3 or 4.
- Regimen B: Febuxostat XR 80 mg Formulation 2: Febuxostat XR 80 mg capsule formulation 2 (F2), orally, once on Day 1 of periods 1, 2, 3 or 4.
- Regimen C: Febuxostat XR 80 mg Formulation 3: Febuxostat XR 80 mg capsule formulation 3 (F3), orally, once on Day 1 of periods 1, 2, 3 or 4.
- Regimen D: Febuxostat XR 80 mg Formulation 4: Febuxostat XR 80 mg capsule formulation 4 (F4), orally, once on Day 1 of periods 1, 2, 3 or 4.
Arm/Group | Regimen A: Febuxostat XR 80 mg Formulation 1 | Regimen B: Febuxostat XR 80 mg Formulation 2 | Regimen C: Febuxostat XR 80 mg Formulation 3 | Regimen D: Febuxostat XR 80 mg Formulation 4
Number analyzed (Participants) | 76 | 74 | 77 | 76
ng/mL | 2027.1184 (1278.28368) | 1442.2267 (991.94583) | 1730.2468 (1013.56204) | 1809.3158 (1170.53245)
Statistical Analysis 1: Comparison: Regimen A: Febuxostat XR 80 mg Formulation 1 vs Regimen D: Febuxostat XR 80 mg Formulation 4; Relative bioavailability of a single dose of Febuxostat XR 80 mg in test (Regimen A) and reference (Regimen D); Test type: Non-Inferiority or Equivalence — Bioequivalence of Febuxostat formulation 1, 2, and 3 to Febuxostat formulation 4 was declared if the 90% confidence intervals for the ratios of central values were within the pre-specified interval of 0.80 to 1.25; Point Estimate = 1.0848, 90% CI 2-sided [0.9528 to 1.2350] — Point estimate and 90% CI were obtained from the exponentiated results of analysis of the natural log (ln)-transformed parameters was performed with regimen, sequence, period, and participants nested within sequence as fixed effects
Statistical Analysis 2: Comparison: Regimen B: Febuxostat XR 80 mg Formulation 2 vs Regimen D: Febuxostat XR 80 mg Formulation 4; Relative bioavailability of a single dose of Febuxostat XR 80 mg in test (Regimen B) and reference (Regimen D); Test type: Non-Inferiority or Equivalence — [test comment as in outcome 1, analysis 1]; Point Estimate = 0.7709, 90% CI 2-sided [0.6767 to 0.8782] — [estimate comment as in outcome 1, analysis 1]
Statistical Analysis 3: Comparison: Regimen C: Febuxostat XR 80 mg Formulation 3 vs Regimen D: Febuxostat XR 80 mg Formulation 4; Relative bioavailability of a single dose of Febuxostat XR 80 mg in test (Regimen C) and reference (Regimen D); Test type: Non-Inferiority or Equivalence — [test comment as in outcome 1, analysis 1]; Point Estimate = 0.9389, 90% CI 2-sided [0.8246 to 1.0689] — [estimate comment as in outcome 1, analysis 1]

2. Primary Outcome: Mean AUCt: Area Under the Plasma Concentration-Time Curve From Time 0 to the Time of the Last Quantifiable Concentration for Febuxostat
Description: AUCt is a measure of total plasma exposure to the drug from time 0 to time of the last quantifiable concentration.
Time Frame: Day 1 pre-dose and at multiple time points (up to 48 hours) post-dose
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: ng*hr/mL
Arm/Group | Regimen A: Febuxostat XR 80 mg Formulation 1 | Regimen B: Febuxostat XR 80 mg Formulation 2 | Regimen C: Febuxostat XR 80 mg Formulation 3 | Regimen D: Febuxostat XR 80 mg Formulation 4
Number analyzed (Participants) | 76 | 75 | 77 | 76
ng*hr/mL | 9395.6014 (3961.55203) | 7971.0624 (3291.36390) | 8652.7080 (3673.91666) | 8817.3600 (3429.94880)
Statistical Analysis 1: Comparison: Regimen A: Febuxostat XR 80 mg Formulation 1 vs Regimen D: Febuxostat XR 80 mg Formulation 4; Relative bioavailability of a single dose of Febuxostat XR 80 mg in test (Regimen A) and reference (Regimen D); Test type: Non-Inferiority or Equivalence — [test comment as in outcome 1, analysis 1]; Point Estimate = 1.0435, 90% CI 2-sided [0.9840 to 1.1066] — [estimate comment as in outcome 1, analysis 1]
Statistical Analysis 2: Comparison: Regimen B: Febuxostat XR 80 mg Formulation 2 vs Regimen D: Febuxostat XR 80 mg Formulation 4; Relative bioavailability of a single dose of Febuxostat XR 80 mg in test (Regimen B) and reference (Regimen D); Test type: Non-Inferiority or Equivalence — [test comment as in outcome 1, analysis 1]; Point Estimate = 0.8777, 90% CI 2-sided [0.8274 to 0.9311] — [estimate comment as in outcome 1, analysis 1]
Statistical Analysis 3: Comparison: Regimen C: Febuxostat XR 80 mg Formulation 3 vs Regimen D: Febuxostat XR 80 mg Formulation 4; Relative bioavailability of a single dose of Febuxostat XR 80 mg in test (Regimen A) and reference (Regimen D); Test type: Non-Inferiority or Equivalence — [test comment as in outcome 1, analysis 1]; Point Estimate = 0.9540, 90% CI 2-sided [0.8996 to 1.0117] — [estimate comment as in outcome 1, analysis 1]

3. Primary Outcome: Mean AUC∞: Area Under the Plasma Concentration-time Curve From Time 0 to Infinity for Febuxostat
Description: AUC∞ is a measure of total plasma exposure to the drug from time zero extrapolated to infinity.
Time Frame: Day 1 pre-dose and at multiple time points (up to 48 hours) post-dose
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: ng*hr/mL
Arm/Group | Regimen A: Febuxostat XR 80 mg Formulation 1 | Regimen B: Febuxostat XR 80 mg Formulation 2 | Regimen C: Febuxostat XR 80 mg Formulation 3 | Regimen D: Febuxostat XR 80 mg Formulation 4
Number analyzed (Participants) | 69 | 62 | 69 | 69
ng*hr/mL | 9368.0744 (3944.01280) | 8278.6143 (3205.31556) | 8938.8765 (3746.60153) | 9102.3700 (3430.45699)
Statistical Analysis 1: Comparison: Regimen A: Febuxostat XR 80 mg Formulation 1 vs Regimen D: Febuxostat XR 80 mg Formulation 4; Relative bioavailability of a single dose of Febuxostat XR 80 mg in test (Regimen A) and reference (Regimen D); Test type: Non-Inferiority or Equivalence — [test comment as in outcome 1, analysis 1]; Point Estimate = 1.0283, 90% CI 2-sided [0.9691 to 1.0911] — [estimate comment as in outcome 1, analysis 1]
Statistical Analysis 2: Comparison: Regimen B: Febuxostat XR 80 mg Formulation 2 vs Regimen D: Febuxostat XR 80 mg Formulation 4; Relative bioavailability of a single dose of Febuxostat XR 80 mg in test (Regimen B) and reference (Regimen D); Test type: Non-Inferiority or Equivalence — [test comment as in outcome 1, analysis 1]; Point Estimate = 0.9056, 90% CI 2-sided [0.8516 to 0.9630] — [estimate comment as in outcome 1, analysis 1]
Statistical Analysis 3: Comparison: Regimen C: Febuxostat XR 80 mg Formulation 3 vs Regimen D: Febuxostat XR 80 mg Formulation 4; Relative bioavailability of a single dose of Febuxostat XR 80 mg in test (Regimen C) and reference (Regimen D); Test type: Non-Inferiority or Equivalence — [test comment as in outcome 1, analysis 1]; Point Estimates = 0.9463, 90% CI 2-sided [0.8909 to 1.0051] — [estimate comment as in outcome 1, analysis 1]

ADVERSE EVENTS:
Time Frame: From the first administration of study drug on Day 1 of Period 1 up to 30 days after the last dose of study drug or Early termination visit (approximately up to 95 days)
Description: At each visit the investigator had to document any occurrence of adverse events and abnormal laboratory findings. Any event spontaneously reported by the participant or observed by the investigator was recorded, irrespective of the relation to study treatment. Safety Set included all participants who received at least 1 dose of study drug.
Arm/Group | Regimen A: Febuxostat XR 80 mg Formulation 1 | Regimen B: Febuxostat XR 80 mg Formulation 2 | Regimen C: Febuxostat XR 80 mg Formulation 3 | Regimen D: Febuxostat XR 80 mg Formulation 4
Serious Adverse Events (participants affected / at risk) | 0/76 | 1/76 | 0/77 | 0/76
Other Adverse Events (participants affected / at risk) | 6/76 | 9/76 | 7/77 | 7/76
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Regimen A: Febuxostat XR 80 mg Formulation 1 (N=76) | Regimen B: Febuxostat XR 80 mg Formulation 2 (N=76) | Regimen C: Febuxostat XR 80 mg Formulation 3 (N=77) | Regimen D: Febuxostat XR 80 mg Formulation 4 (N=76)
Blood creatine phosphokinase increased (Investigations) | 0 | 1 | 0 | 0
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Regimen A: Febuxostat XR 80 mg Formulation 1 (N=76) | Regimen B: Febuxostat XR 80 mg Formulation 2 (N=76) | Regimen C: Febuxostat XR 80 mg Formulation 3 (N=77) | Regimen D: Febuxostat XR 80 mg Formulation 4 (N=76)
Diarrhoea (Gastrointestinal disorders) | 0 | 0 | 2 | 0
Nausea (Gastrointestinal disorders) | 1 | 0 | 0 | 1
Vomiting (Gastrointestinal disorders) | 0 | 1 | 0 | 0
Nasopharyngitis (Infections and infestations) | 0 | 2 | 0 | 0
Bacterial vaginosis (Infections and infestations) | 1 | 0 | 0 | 0
Oral herpes (Infections and infestations) | 0 | 0 | 0 | 1
Trichomoniasis (Infections and infestations) | 0 | 1 | 0 | 0
Contusion (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 1
Back pain (Musculoskeletal and connective tissue disorders) | 1 | 1 | 0 | 0
Myalgia (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0 | 0
Headache (Nervous system disorders) | 1 | 2 | 1 | 3
Syncope (Nervous system disorders) | 1 | 0 | 1 | 0
Dizziness (Nervous system disorders) | 0 | 1 | 0 | 0
Presyncope (Nervous system disorders) | 0 | 0 | 1 | 0
Libido decreased (Psychiatric disorders) | 0 | 0 | 1 | 0
Dysmenorrhoea (Reproductive system and breast disorders) | 0 | 1 | 0 | 0
Vaginal discharge (Reproductive system and breast disorders) | 0 | 1 | 0 | 0
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 | 0
Dry skin (Skin and subcutaneous tissue disorders) | 0 | 1 | 0 | 0
Papule (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 1
Pruritus (Skin and subcutaneous tissue disorders) | 0 | 0 | 1 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Research Organization shall not publish any articles or papers nor make any presentations, nor assist any other person in publishing any articles or papers or in making any presentations relating or referring to the Study or any results, data or insights from or any data, information or materials obtained or generated in the performance of its obligations without the prior written consent of Takeda, which consent may be granted or withheld in Takeda's sole discretion.